CLINICAL TRIAL: NCT03903432
Title: The Feasibility of Using MRI During Endoscopic Sinus Surgery
Brief Title: The Feasibility of Using MRI During ESS
Acronym: ESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roee Landsberg (Other)
Collaborators: Assuta Medical Center (Other)
Responsible Party: Sponsor-Investigator, Roee Landsberg, Principal Investigator, Assuta Medical Center
Organization: Assuta Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0059-18-ASMC
Record Dates: First submitted 2019-01-30; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Chronic Sinusitis
Keywords: MRI; CT; Chronic Sinusitis; ESS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 45 participants, in one center - Assuta (Other): Patients with chronic sinusitis who are scheduled to undergo ESS at Assuta will be recruited and patients will sign an informed consent form for performing MRI (new protocol-without gadolinium injection) in addition to the routine CT.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — candidates for ESS will be referred to conventional CT scans of the sinuses. If surgery is to be performed, the patients will sign an informed consent and be referred for a sinus MRI.
  Other Names: CT

SUMMARY:
Before performing endoscopic sinus surgery (ESS-Endoscopic Sinus Surgery), every candidate for surgery is referred to perform a sinus CT scan of the sinuses. Because of the complicated anatomy of the sinuses and their proximity to vital organs such as the brain, eye, and carotid artery, the surgeon use the CT imaging during surgery to adjust the anatomy and to avoid complications such as blindness, brain damage and massive bleeding (0.3%). Sometimes the CT is integrated into a navigation system, although there is no evidence that the use of navigation systems reduces the rate of complications.

The aim of our study is to examine whether ESS can be performed in chronic sinusitis patients using MRI, with CT being used as a backup only.

DETAILED DESCRIPTION:
The sinuses are different from person to person and from side to side, and therefore it is essential to be completely familiar with the anatomy of the specific patient.

The sinuses are a maze of cells filled with air and surrounded by thin bony partitions separating the cells, as well as separating the nasal and sinus cavities from the vital organs mentioned.

CT imaging is the standard test because it allows accurate detection of the bony partitions, thus contributing to the accuracy and safety of the operation.

The known disadvantage of the CT is its radiation. The amount of radiation is not negligible and involves the possible development of eye damage (cataracts) or tumors.

For a large number of patients, the CT imaging performed before surgery is neither the first nor the last, so that the risk of tumor disease increases significantly, especially for the younger population. Another disadvantage is the limited ability of the imaging to demonstrate soft tissue.

Compared to CT, MRI is better for soft tissue demonstration. Another important advantage is that it is a radiation-free scan. Its disadvantages are a poor demonstration of the bony partitions and being relatively long, expensive, and therefore less available.

Although the CT is more accurate in demonstrating bony structures, cheaper and more accessible, the radiation risk is very disturbing to both the physicians and patients who have become more aware of the problem in recent years.

Among neurosurgeons, whose field of operation is very close to the surgical field of sinus surgeons (for example, in the trans-sphenoidal surgery of the pituitary gland), surgery is often performed only with MRI.

When a potential patient arrives for sinus surgery with an MRI, some sinus surgeons will skip the CT. However, this practice does not yet have an orderly basis, and that is where the investigators are aiming.

In a previous study, the initiators (rhinologist and neuroradiologist) suggested that MRI parameters could be upgraded to allow a better and clearer demonstration of the bony partitions, so that the surgeon could rely on the anatomy derived from this scan. As a result of the desired change, the patients will not be exposed to radiation, and at the same time, a better demonstration of the soft tissues will also be possible.

In this study, 20 patients who performed CT imaging prior to ESS were sent to perform sinus MRI (new protocol- without gadolinium injection). Twenty-three bony anatomical structures were selected that are important for the surgeon's orientation. The rhinologist and neuroradiologist independently evaluated the CT and MRI of each patient and compared it by giving a numerical score for the degree of visibility of each structure.

In both disciplines, in about 55% of cases, the structures observed in MRI were observed similarly in CT. According to the rhinologist, in 84% the CT was similar or better. According to the neuroradiologist, in 86% the MRI was similar or better. Still, even for the rhinologist, in 67% the MRI was similar or better.

Therefore, according to this protocol, it was found that in both disciplines, most of the anatomical structures are well observed on MRI.

adding the obvious superiority of MRI over CT in soft tissue demonstration, the investigators conclude that MRI use in ESS can be considered at least in some cases.

the investigators assume that a neuroradiologist has an advantage in reading MRI, and that an rhinologist has an advantage in reading CT. It should be expected that over time and after a learning curve, MRI readings among rhinologist will improve. This study is about to be published these days.

Encouraged by its results, it is now necessary to examine the feasibility of the conclusions in real setting.

Endpoints:

1. Statistics will be carried out for all 15 questionnaires of each surgeon on questions a-g:

   1. The level of surgery using MRI
   2. Safety level using MRI
   3. Use of CT during surgery
   4. Continuous work with MRI
   5. Ease of work in different sinus groups
   6. Complications when working with MRI
   7. Would the surgeon's exposure to CT imaging change the operation?
2. Statistics will be carried out for all 15 questionnaires of each surgeon on questions a-b.

   1. Would the surgeons prefer to work with MRI instead of CT?
   2. Scoring of the following diseases according to the convenience of working with the MRI scan: 1-comfortable, 2-medium, 3-uncomfortable.

      1. Chronic sinusitis with polyposis (1-2-3)
      2. Chronic sinusitis without polyposis (1-2-3)
      3. Antrochoanal polyp (1-2-3)
      4. Fungal ball (1-2-3)
      5. Allergic fungal sinusitis (1-2-3)
      6. Sinus mucocele (1-2-3)
      7. Odontogenic sinusitis (1-2-3)
      8. Deviated nasal septum (1-2-3)
      9. Inferior turbinates hypertrophy (1-2-3)
3. Comparative statistics of all the above will be carried out between the average of the questions of the three surgeons.

Number of participants, and number of centers planned to participate in the study:

45 participants, in one center - Assuta

Methods/ protocol:

* Three sinus surgeons will be selected.
* Each surgeon will recruit 15 patients for the study, a total of 45 patients.
* Follow-up patients who are potential candidates for ESS will be referred to conventional CT scans of the sinuses.
* The surgeons will be exposed to the verbal interpretation of the scan, in order to finally decide whether to operate or not, but not to the imaging itself.
* If surgery is to be performed, the patients will sign an informed consent and be referred for a sinus MRI.
* Before surgery, the surgeon will not look at the CT imaging, but only on MRI.
* Prior to surgery, the surgeons will be instructed about the new MRI protocol by the neuroradiologist.
* The operation will be performed when only the MRI is displayed on the screen. However, the CT scan will also be in the operating room in case the surgeon feels that the MRI is insufficient.
* The surgeons will observe the CT scan after the surgery, and then complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic sinusitis.
2. Patients designated for ESS surgery.

Exclusion Criteria:

1. Patients who have already undergone ESS and/ or nasal septum/ turbinates surgery.
2. Patients with sinus cancer.
3. Patients after sinus injury.
4. Patients under 18 years of age.
5. Extreme Situations: The radiologist who analyzes the CT and MRI will warn of situations in which he or she will detect an increased risk of injury to vital organs.

These situations will include:

A. Dehiscence, as seen in CT, in the bony walls of:

1. The carotid artery.
2. Skull base.
3. Medial wall of the orbit.

B. Situations in which an anatomical anomaly or distortion of the nasal or sinus cavity is observed in the CT imaging.

C. Situations in which the radiologist identifies poor technical quality of the MRI, and, in particular, a poor demonstration of the bony components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Ease and saftey of use of MRI compared to CT during ESS | imediatly after surgery is done (+- 12 hours)
  A questionnaire to assess the feasibility and ease of use of MRI during surgery will be filled out by the surgeon at the end of each surgery.
  1. What was your general feeling about this surgery using MRI as compared to a similar surgery in which you used CT? A SCALE OF 1-2-3 where 1- BETTER 2- SAME 3- WORSE
  2. Safety level using MRI compared to CT? A SCALE OF 1-2-3 where 1- BETTER 2- SAME 3- WORSE
  3. please rate the level of Ease of work in the different sinus groups (on a scale of 1-2-3 where 1- easy 2- somewhat easy 3- not easy)
the impact of using MRI compared to CT during ESS Ease and saftey of use of MRI compared to CT during ESS | imediatly after surgery is done (+- 12 hours)
  A questionnaire to assess the feasibility and ease of use of MRI during surgery will be filled out by the surgeon at the end of each surgery.
  1. How many times was there a sporadic Use of CT during surgery (1-3 times)? (yes / no)
  2. Was there a need for Continuous work with CT? (yes / no)
  3. were there any complications when working with MRI ( no / yes, if yes please elaborate)
  4. Do you think that an exposure to CT imaging would have changed the operation? If yes please elaborate

CONTACTS AND LOCATIONS:
Overall Officials: Roee Landsberg, M.D, Principal Investigator — Assuta Hospital 1st Floor Habarzel Street 20 Ramat Hahayal Tel Aviv
Locations (1):
- Assuta Hospital 1st Floor Habarzel Street 20 Ramat Hahayal Tel Aviv, Tel Aviv, Israel